CLINICAL TRIAL: NCT03705468
Title: Assessment of Kétamine and Propofol Sedation During Intra Tracheal Surfactant Administration by the LISA Method (Less Invasive Surfactant Administration)
Brief Title: Assessment of Ketamine and Propofol Sedation During LISA Method (Less Invasive Surfactant Administration)
Acronym: ANALISA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0340
Record Dates: First submitted 2018-09-04; First posted 2018-10-15 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Premature Neonate
Keywords: Less Invasive Surfactant Administration (LISA); Sedation; RDS treated by CPAP requiring surfactant; Sedation during intra tracheal surfactant administration by the LISA method; Available intravenous line
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ketamine sedation: Ketamine sedation
- Propofol sedation: Propofol sedation

SUMMARY:
Respiratory distress syndrome (RDS) caused by surfactant deficiency remains one of the major reasons of morbi-mortality in preterm infants and affects 85% of preterm babies born less than 32 week gestational age (wGA). The strategy to manage RDS relies on the use of surfactant and non-invasive nasal ventilation, to limit tracheal mechanical ventilation. During recent years, surfactant administration through a thin catheter in spontaneously breathing preterm used in association with continuous positive airway pressure (CPAP) has emerged as a new approach for treating neonates with respiratory failure. The main objectives of Less Invasive Surfactant Administration (LISA) are to avoid endotracheal mechanical ventilation and its side effects including bronchopulmonary dysplasia. The LISA premedication procedure still under debate, because only 1 trial use analgesia or sedation during procedure. This reflects neonatologists concerns about side effects (apnea and the need for mechanical ventilation) of this premedication. This study aims to optimize sedation during LISA procedure by evaluating pain score with Ketamine or Protofol sedation, in Neonatal intensive care unit (NICU) patients with RDS.

DETAILED DESCRIPTION:
Systematic reviews of the prospective studies performed suggest that among preterm infants, the use of LISA was associated with the lowest likelihood of the composite outcome of death or bronchopulmonary dysplasia (BPD) at 36 weeks' postmenstrual age when compared with the other ventilation strategies for preterm infants. Further studies are needed to optimize the indications and identify adequate strategies for premedication that preserve respiratory function and which limits pain and cardio-respiratory instability associated with laryngeal exposure without increasing risks of complications. According to a recent European survey, only 48% of neonatologists perform LISA with sedation. In a recent retrospective study, Dekker showed a more favorable COMFORTneo score with Propofol versus without, similar rates of intubation during LISA. Ketamine infusion has been used in several NICUs with few reported effects on respiratory function, but without publication. No prospective studies exist on LISA premedication. This study aims to optimize sedation during LISA in NICU patients with RDS. Comparing Ketamine and propofol sedation with rate of mechanical tracheal ventilation from the start of the LISA procedure up to 2 hours of life, in the NICU of Arnaud de Villeneuve University Hospital of Montpellier (France).

ELIGIBILITY:
Inclusion Criteria:

* Infant born below 30 wGA with RDS treated by CPAP requiring surfactant
* Available IV line
* Admission to the NICU of Montpellier University Hospital Centre in the first 24 hours of life

Exclusion Criteria:

* maternal general anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infant born below 30 wGA with RDS treated by CPAP requiring surfactant and Available IV line
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Rate of mechanical ventilation (MV) from the start of the LISA procedure up to 2 hours of life | 2 hours after LISA procedure
  The Investigators would like to evaluating the need for MV within the time of the LISA procedure and up to 2 hours of life among preterm babies less than 30wGA

SECONDARY OUTCOMES:
Cardiorespiratory parameters | 5 and 30 minutes after the drug injection 24 and 72 hours of life and 36 week gestational age
  Cardiorespiratory parameters before and at 5, 30 minutes after the drug injection: blood pressure
Cardiorespiratory parameters | 5 and 30 minutes after the drug injection 24 and 72 hours of life and 36 week gestational age
  Cardiorespiratory parameters before and at 5, 30 minutes after the drug injection: FiO2
Cardiorespiratory parameters | 5 and 30 minutes after the drug injection 24 and 72 hours of life and 36 week gestational age
  Cardiorespiratory parameters before and at 5, 30 minutes after the drug injection: heart rate
Rate of MV from the start of the LISA procedure up to 24 and 72 hours of life and causes of failure | 5 and 30 minutes after the drug injection 24 and 72 hours of life and 36 week gestational age
  Rate of MV from the start of the LISA procedure up to 24 and 72 hours of life and causes of failure (apnea, need surfactant)
To assess Neonatal morbidity at 36 wGA | 5 and 30 minutes after the drug injection 24 and 72 hours of life and 36 week gestational age
  Neonatal morbidity at 36 wGA
To assess mortality at 36 wGA | 5 and 30 minutes after the drug injection 24 and 72 hours of life and 36 week gestational age
  Mortality at 36 wGA

CONTACTS AND LOCATIONS:
Overall Officials: MILESI Christophe, PUPH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

REFERENCES:
- [Derived] Brotelande C, Milesi C, Combes C, Durand S, Badr M, Cambonie G. Premedication with ketamine or propofol for less invasive surfactant administration (LISA): observational study in the delivery room. Eur J Pediatr. 2021 Sep;180(9):3053-3058. doi: 10.1007/s00431-021-04103-1. Epub 2021 May 6. PMID 33954805